CLINICAL TRIAL: NCT03725865
Title: A Clinical Study of Intracerebral Transplantation of Human Peripheral Blood Derived Induced Neural Stem Cells for Cerebral Hemorrhagic Stroke
Brief Title: A Clinical Study of iNSC Intervent Cerebral Hemorrhagic Stroke
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iNSC-81NK-01
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iNSC treatment group (Experimental)
  Interventions: Biological: Induction of neural stem cells

INTERVENTIONS:
Biological: Induction of neural stem cells — Brain injection iNSC

SUMMARY:
This is a single centre、single arm、open-label，to investigate the safety and efficacy of induction of neural stem cells transplantation in the brain

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, provide written informed consent, and comply with the study procedures.
2. Men and women 30-65 years old.
3. Women must have a negative serum pregnancy test, gestation age women practice an acceptable method of contraception.
4. At least 12 months but no more than 60 months from time of hemorrhagic stroke, with a motor neurological deficit.
5. Documented history of single hemorrhagic stroke in subcortical region of MCA or lenticulostriate artery with or without cortical involvement, with correlated findings by MRI.
6. Modified Rankin Score of 2, 3 or 4.
7. FMMS score of 55 or less, two evaluations at approximately 3 weeks apart prior to surgery with less than +/- 5 point change in the FMMS.
8. Two evaluations at approximately 3 weeks apart prior to surgery with less than +/- 4 point change in the NIHSS.
9. Able and willing to undergo post-physical therapy/rehabilitation.

Exclusion Criteria:

1. Any disabling psychological or psychiatric disorders which may confound the study.
2. History of more than one hemorrhagic stroke.
3. History of another major neurological disease or injury.
4. Cerebral soften lesion size >5cm in any one measurement.
5. Myocardial infarction within the prior 3 months.
6. History of seizures or current use of antiepileptic medication.
7. History of peripheral nerve surgery, including Selective Dorsal Rhizotomy and Contralateral Seventh Cervical Nerve Transfer.
8. Receipt of any investigational drug or device within 30 days.
9. Receipt of any cell infusion other than blood transfusion.
10. Any concomitant medical disease or condition noted below:

    1. Coagulopathy.
    2. Active or history of malignancy.
    3. Primary or secondary immune deficiency.
    4. Persistent MRI artifact or unable to undergo MRI.
11. Any condition that the Investigator or primary physician feels may interfere with participation in the study or may endanger the subject.
12. Any condition that the surgeon feels may pose complications for the surgery.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent AE | 1 year